CLINICAL TRIAL: NCT00417274
Title: An Open-Label, Phase II Safety, Tolerability, Drug Level and Efficacy Trial of Quinacrine in Patients With Androgen-Independent Metastatic Prostate Cancer
Brief Title: Quinacrine Treatment in Patients With Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cleveland BioLabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBL-DD-05-C-H-2003
Record Dates: First submitted 2006-12-27; First posted 2006-12-29 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2012-09

CONDITIONS: Prostatic Cancer
Keywords: Cancer of Prostate; Prostate Cancer; Cancer of the Prostate; Neoplasms, Prostate; Neoplasms, Prostatic; Prostate Neoplasms; Prostatic Cancer; Androgen-Independent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Quinacrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quinacrine (Experimental): Uncontrolled treatment arm
  Interventions: Drug: Quinacrine

INTERVENTIONS:
Drug: Quinacrine — 100 mg daily
  Other Names: CBLB102

SUMMARY:
The purpose of this study is to determine whether quinacrine is effective in the treatment of Androgen-Independent Prostate Cancer.

DETAILED DESCRIPTION:
Despite a modest improvement in survival with available chemotherapy treatments, androgen-independent metastatic prostate cancer remains essentially incurable.

Several changes in gene function that characterize malignancy have been identified. For example the p53 gene in normal tissue lessens the risk of cancer through growth arrest or cell suicidal programs. Thus the silenced p53 gene present in cancer tissue contributes to the growth of the cancer. In addition when the p53 gene is silenced, a cell survival pathway, controlled by the NF-kB gene, is activated leading increased cell survival.

Quinacrine can activate p53 and inhibit NF-kB, thus reestablishing cell suicidal programs and decreasing cell survival in cancer tissue. Moreover, quinacrine is effective against several prostate tumor cell lines in vitro, and has anti-tumor effects against prostate cancer xenografts in mice.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be males, at least 18 years of age, with pathologically confirmed adenocarcinoma of the prostate
* Patients must have evidence of androgen-independent metastatic prostate cancer (AIMPC) following standard antiandrogen withdrawal. AIMPC will be defined as the category of patients with metastatic prostate cancer with radiologic evidence of metastases (bone scan, CT, etc.) and castrate levels of testosterone (~ 50 ng/dL).

  1. All patients must be receiving ongoing therapy to ensure testicular androgen suppression (LHRH agonists therapy or bilateral orchiectomy).
  2. All patients receiving anti-androgen therapy [e.g., flutamide (Eulexin), bicalutamide (Casodex), or nilutamide (Nilandron)] must have initiated therapy at least 3 months (90 days) prior to the Baseline visit.
* Patients must have received prior docetaxel-based or mitoxantrone-based chemotherapy, or refused or been ineligible for chemotherapy. Previous chemotherapy treatments must be completed at least 4 week prior to Screening, and patients must not have any residual therapy-related toxicities present at Screening.
* Patients must have evidence of disease progression defined as any of the following:

  1. New sites of metastatic disease on radiographic imaging (bone scan or CT scan of chest/abdomen/pelvis) as determined by the referring physician.
  2. PSA progression, defined as a 50% or greater rise in PSA value over a baseline level of at least 1.0 ng/mL, confirmed after an interval of at least two weeks.
* ECOG performance status 0-2 (see Appendix 4)
* Patients must have adequate organ and bone marrow function as defined below:

  1. Absolute neutrophil count greater than 1500/mL
  2. Platelets greater than 100,000/mL
  3. Serum creatinine less than 2.0 mg/dL
  4. Total bilirubin less than 1.5 mg/dL
  5. AST (SGOT) and ALT (SGPT) less than 2 times the ULN [less than 5 times the ULN if liver metastases are present].
* Sexually active men whose sexual partners are women of childbearing potential must agree to use a medically acceptable form of barrier contraception or abstinence during their participation in the study and for at least six weeks after study drug discontinuation.
* Written informed consent/HIPAA authorization must be provided prior to the performance of any study-related procedures.

Exclusion Criteria:

* Prior allergic reactions or a history of intolerance attributed to quinacrine or other acridine derivatives
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hematological disorders, hepatic disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Lifetime history of porphyria or psoriasis
* Documented glucose-6-phosphate dehydrogenase deficiency
* Lifetime history of seizure disorder (except infant febrile seizures)
* Lifetime history of schizophrenia, bipolar disorder, or any other psychotic disorders.
* Lifetime history of dermatitis as an allergic/toxic reaction to any medication
* Clinical evidence of CNS metastases
* Patients with a history of any malignancy (other than basal, squamous cell cancers and Ta bladder cancers) within 5 years of baseline visit
* Any grade 2 sensory neuropathy
* QTc (Bazett) >450 msec
* Patients with NYHA class 3 or 4 failure
* Patients with myocardial infarction or acute coronary syndrome within the previous 6 months
* Patients who require anti-arrhythmic treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, MD, Principal Investigator — University of Chicago Hospitals

REFERENCES:
- [Background] Gurova KV, Hill JE, Guo C, Prokvolit A, Burdelya LG, Samoylova E, Khodyakova AV, Ganapathi R, Ganapathi M, Tararova ND, Bosykh D, Lvovskiy D, Webb TR, Stark GR, Gudkov AV. Small molecules that reactivate p53 in renal cell carcinoma reveal a NF-kappaB-dependent mechanism of p53 suppression in tumors. Proc Natl Acad Sci U S A. 2005 Nov 29;102(48):17448-53. doi: 10.1073/pnas.0508888102. Epub 2005 Nov 15. PMID 16287968

RESULTS

PARTICIPANT FLOW:
Groups:
- Quinacrine Treatment: 100 mg once a day
Period: Overall Study
Arm/Group | Quinacrine Treatment
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Quinacrine Treatment: Uncontrolled treatment arm
Arm/Group | Quinacrine Treatment
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Quinacrine, Based on Prostate Specific Antigen (PSA) Response in Patients With Androgen-independent Metastatic Prostate Cancer
Description: Patients who achieved a complete response (CR) or a partial response (PR) to therapy were allowed to continue to receive treatment until disease progression or unacceptable toxicity occurred, until the patient discontinued treatment for another reason, or for a total of 6 months. Patients who continued to show a CR or PR or who maintained stable disease (SD) after 6 months of therapy were to be allowed to continue therapy at the investigator's discretion.
Time Frame: End of treatment
Population: Based on clinical judgment
Measure: Number; unit: Participants
Arm/Group | Quinacrine Treatment
Number analyzed (Participants) | 31
Participants | 1

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Quinacrine Treatment
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinacrine Treatment (N=31)
Thrombosis (Vascular disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
Back pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinacrine Treatment (N=31)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 7 (7)
Electrocardiogram QTc interval prolonged (Cardiac disorders) | 2 (2)
Fatigue (General disorders) | 11 (11)
Fever (General disorders) | 2 (2)
Insomnia (General disorders) | 2 (2)
Weight loss (General disorders) | 7 (7)
Skin disorder (Skin and subcutaneous tissue disorders) | 9 (9)
anorexia (Gastrointestinal disorders) | 9 (9)
constipation (Gastrointestinal disorders) | 5 (5)
diarrhea (Gastrointestinal disorders) | 2 (2)
mucositis (Gastrointestinal disorders) | 2 (2)
taste alteration (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 9 (9)
edema limbs (Blood and lymphatic system disorders) | 6 (6)
Alkaline phosphatse increased (Investigations) | 7 (7)
creatinine increased (Investigations) | 4 (4)
Hyperglycemia (Investigations) | 6 (6)
hypoalbuminemia (Investigations) | 2 (2)
joint disorder (Musculoskeletal and connective tissue disorders) | 3 (3)
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
dizziness (Nervous system disorders) | 5 (5)
back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
headache (Nervous system disorders) | 5 (5)
pain (General disorders) | 12 (12)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
urogenital disorder (Renal and urinary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less